CLINICAL TRIAL: NCT06306222
Title: Comparing the Efficacy of Thulium Fiber Laser vs. Holmium:YAG Laser for the Ureteroscopic Treatment of Patients With Urinary Stone Disease: a Randomized Controlled Trial
Brief Title: Thulium Fiber Laser vs. Holmium:YAG Laser for the Ureteroscopic Treatment of Patients With Urinary Stone Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Eugenio Ventimiglia, Principal investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GR-2021-12375430
Record Dates: First submitted 2023-12-29; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Kidney Stone; Ureteral Stone
MeSH Terms: conditions — Kidney Calculi; Ureterolithiasis | interventions — Lithotripsy, Laser

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thulium fiber laser (TFL) lithotripsy (Experimental): Lithotripsy with TFL is a recently introduced procedure, that will be tested in this study.
  Interventions: Device: Laser lithotripsy
- Holmium:YAG laser lithotripsy (Active Comparator): Holmium:YAG laser lithotripsy represents the gold standard for this procedure since 30 years.
  Interventions: Device: Laser lithotripsy

INTERVENTIONS:
Device: Laser lithotripsy — Ureteroscopic laser lithotripsy

SUMMARY:
This is a randomized controlled trial which aims to compare the efficacy and safety of Thulium fiber laser (TFL) and holmium:yttrium-aluminum-garnet (Ho:YAG) laser ablation during the treatment of upper urinary tract stone disease with flexible ureteroscopy, demonstrating clinical superiority of TFL.

ELIGIBILITY:
Inclusion Criteria:

* Renal/ureteral stones > 4 mm

Exclusion Criteria:

* Anatomical abnormalities

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-11-23 (Estimated); Study Completion 2026-02-23 (Estimated)

PRIMARY OUTCOMES:
Lithotripsy speed | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Stone free rate | 3 months after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No